CLINICAL TRIAL: NCT01005966
Title: Clinical Efficacy of Fluoride Toothpastes Using an in Situ Caries Model
Brief Title: In Situ Caries Model of Fluoride Toothpastes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: T3508605
Record Dates: First submitted 2009-10-15; First posted 2009-11-02 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2012-11

CONDITIONS: Caries
Keywords: remineralization; enamel; in situ; fluoride; caries
MeSH Terms: interventions — fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Run in (Other): Placebo
  Interventions: Drug: Placebo
- Sodium Fluoride Toothpaste (Experimental): Sodium fluoride toothpaste
  Interventions: Drug: Sodium Fluoride Toothpaste
- Amine Fluoride Toothpaste (Active Comparator): Amine Fluoride
  Interventions: Drug: Amine Fluoride Toothpaste
- 675ppmf toothpaste (Other): Dose response
  Interventions: Drug: 675 ppmf toothpaste
- Sodium monofluorophosphate/sodium fluoride Toothpaste (Active Comparator): Sodium monofluorophosphate/sodium fluoride Toothpaste
  Interventions: Drug: Sodium monofluorophosphate/Sodium Fluoride Toothpaste
- 0 ppmf toothpaste (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Fluoride Toothpaste — Test product
  Arms: Sodium Fluoride Toothpaste
Drug: Amine Fluoride Toothpaste — Test product
  Arms: Amine Fluoride Toothpaste
Drug: Sodium monofluorophosphate/Sodium Fluoride Toothpaste — test product
  Arms: Sodium monofluorophosphate/sodium fluoride Toothpaste
Drug: Placebo — placebo and washout treatment
  Arms: 0 ppmf toothpaste; Run in
Drug: 675 ppmf toothpaste — dose response
  Arms: 675ppmf toothpaste

SUMMARY:
This study is to evaluate the effect of fluoride dentrifrices on enamel with artificial caries lesions in an in situ model

ELIGIBILITY:
Inclusion Criteria:

* Consent:Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Age:Aged 18 to 80 years inclusive
* Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions
* General Health:Good general health with (in the opinion of the investigator) no clinically significant and/or relevant abnormalities of medical history or oral examination that could interfere with subject safety during the study period
* Residency: Currently living in the Indianapolis, Indiana area
* Dentures: a) Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accommodate two enamel specimens (required dimensions 12 x 7 millimeters (mm). b) Willing and capable of wearing their removable partial dentures 24 hours per day during each two week treatment period. c) All restorations in a good state of repair
* Salivary Flow: Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/minute; gum base stimulated whole saliva flow rate ≥ 0.8 mL/minute).

Exclusion Criteria:

* Pregnancy:Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Breast-feeding: Women who are breast-feeding
* Allergy/Intolerance:Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Clinical Study/Experimental Medication: a. Participation in another clinical study or receipt of an investigational drug within 30 days of the first treatment visit, with the exception of study GSK dental studies where the wash in period prior to treatment is sufficient. b. Previous participation in this study
* Antibiotics: Currently taking antibiotics or have taken antibiotics in the two weeks prior to the screening visit
* Fluoride: Prescribed or professionally recommended use of fluoride supplements or fluoride mouthrinse
* Substance abuse: Recent history (within last year) of alcohol or other substance abuse
* Dental Health: Current active caries or periodontal disease that may compromise the study or health of the subjects
* Personnel: a. A member of the site study staff who is directly working on the project or living in that staff's household. b. An employee of the sponsor c. Any employee of any toothpaste manufacturer or their spouse or family member

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: 83 participants were screened and 18 participants did not meet the study criteria thus 65 participants were enrolled into the study. The subjects were randomized to receive all 5 study treatments in a pre-determined computerized randomised order as per a typical cross-over design.
Groups:
- Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F]: Study toothpaste containing sodium fluoride/ silica (1426ppm fluoride as NaF)
- Amine Fluoride(AmF) Toothpaste (1400ppmF): Reference toothpaste containing amine fluoride (1400ppm fluoride as AmF)
- Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF): Reference toothpaste containing sodium monofluorophosphate and sodium fluoride (1450ppmF - 1000ppmF as NaMFP and 450ppmF as NaF)
- NaF Toothpaste (675ppmF): Study toothpaste containing sodium fluoride and silica (675ppmF as NaF)
- Placebo Toothpaste (0ppmF): Placebo fluoride free toothpaste
Period: Treatment Period 1 (14 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 13 | 13 | 13 | 13 | 13
Completed | 11 | 13 | 12 | 13 | 13
Not Completed | 2 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0
Period: Washout Period 1 (4 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 11 | 13 | 12 | 13 | 13
Completed | 11 | 13 | 12 | 12 | 13
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Treatment Period 2 (14 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 13 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 13 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 1) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 1)
Completed | 13 | 12 | 10 | 11 | 11
Not Completed | 0 | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Washout Period 2 (4 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 13 | 12 | 10 | 11 | 11
Completed | 13 | 12 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (14 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 8 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 13 (Due to crossover design, a different set of subjects received this treatment compared to Period 2) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 2)
Completed | 12 | 7 | 12 | 13 | 11
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1
Period: Washout Period 3 ( 4 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 12 | 7 | 12 | 13 | 11
Completed | 12 | 7 | 12 | 13 | 11
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4 (14 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 3) | 13 (Due to crossover design, a different set of subjects received this treatment compared to Period 3)
Completed | 10 | 10 | 11 | 10 | 12
Not Completed | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Other Reason | 0 | 0 | 0 | 0 | 1
Period: Washout Period 4 (4 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 10 | 10 | 11 | 10 | 12
Completed | 10 | 10 | 11 | 10 | 12
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5 (14 Days)
Arm/Group | Sodium Fluoride(NaF) Toothpaste[1426parts Per Million(Ppm)F] | Amine Fluoride(AmF) Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 9 (Due to crossover design, a different set of subjects received this treatment compared to Period 4) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 4) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 4) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 4) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 4)
Completed | 9 | 12 | 11 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who received at least one dose of the study treatments or who have been evaluated for AEs were included.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 65
Age Continuous [Mean (Standard Deviation); unit: years] | 67.0 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Percent Surface Microhardness (SMH) Recovery of Enamel Specimens Exposed to NaF Toothpaste (1426ppmF) and AmF Toothpaste (1400ppmF)
Description: SMH recovery test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. Difference in percent SMH recovery was calculated by comparing study NaF toothpaste (1426ppmF) with reference AmF toothpaste (1400ppmF).
Time Frame: Baseline to 14 days
Population: Per protocol (PP) population: All randomized participants who received at least one dose of the study treatments and provided at least one measurement SMH. Participants without any major protocol violations in given study treatment period were included in the PP population.
Measure: Mean (Standard Error); unit: Percentage SMHR
Groups:
- NaF Toothpaste (1426ppmF): Study toothpaste containing NaF/ silica (1426ppmF)
- AmF Toothpaste (1400ppmF): Reference toothpaste containing AmF (1400ppmF)
Arm/Group | NaF Toothpaste (1426ppmF) | AmF Toothpaste (1400ppmF)
Number analyzed (Participants) | 56 | 57
Percentage SMHR | 38.05 (2.52) | 41.06 (2.53)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426ppmF) vs AmF Toothpaste (1400ppmF); Null hypothesis considered population means for NaF toothpaste and AmF toothpaste to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p = 0.2117, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; Analysis of variance (ANOVA) based on a mixed model with the factors subject, treatment and period was used; Adjusted Mean Difference = -3.01, 95% CI 2-sided [-7.75 to 1.73] — Statistical tests were 2-sided with a significance level of 0.05

2. Secondary Outcome: Percent SMH Recovery of Enamel Specimens Exposed to NaF Toothpaste (1426ppmF), NaF Toothpaste (675ppmF), NaMFP/NaF Toothpaste (1400ppm F) and Placebo (0ppmF)
Description: SMH test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. Differences in percent SMH recovery due to study and reference toothpastes were calculated.
Time Frame: Baseline to 14 days
Population: PP population: All randomized participants who received at least one dose of the study treatments or provided at least one measurement SMH. Participants without any major protocol violations in given study treatment period were included in the PP population.
Measure: Mean (Standard Error); unit: Percentage SMHR
Groups:
- AmF Toothpaste (1400ppmF): Reference toothpaste containing AmF(1400ppmF)
- NaMFP/NaF Toothpaste (1450ppmF): Reference toothpaste containing NaMFP/NaF (1450ppmF- 1000ppmF as NaMFP and 450ppmF as NaF)
- NaF Toothpaste (675ppmF): Toothpaste containing NaF/silica (675ppmF)
- Placebo Toothpaste (0ppmF): Placebo - fluoride free toothpaste
Arm/Group | NaF Toothpaste (1426ppmF) | AmF Toothpaste (1400ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Number analyzed (Participants) | 56 | 57 | 58 | 59 | 59
Percentage SMHR | 38.05 (2.52) | 41.06 (2.53) | 33.48 (2.49) | 29.08 (2.50) | 14.49 (2.48)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426ppmF) vs NaF Toothpaste (675ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and NaF toothpaste (675ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p = 0.0002, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 8.96, 95% CI 2-sided [4.27 to 13.66] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 2: Comparison: NaF Toothpaste (1426ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and Na MFP/NaF toothpaste (1450ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p = 0.0557, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 4.57, 95% CI [-0.11 to 9.24] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 3: Comparison: NaF Toothpaste (1426ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and Placebo toothpaste (0ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 23.55, 95% CI 2-sided [18.86 to 28.24] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 4: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); Null hypothesis considered population means for the Na MFP/NaF toothpaste (1450ppmF) and NaF toothpaste (675ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p = 0.0625, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 4.40, 95% CI 2-sided [-0.23 to 9.03] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 5: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for the Na MFP/NaF toothpaste (1450ppmF) and Placebo toothpaste (0ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 18.99, 95% CI 2-sided [14.36 to 23.61] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 6: Comparison: NaF Toothpaste (675ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for the NaF toothpaste (675ppmF) and Placebo toothpaste (0ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 14.59, 95% CI 2-sided [9.95 to 19.23] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 7: Comparison: AmF Toothpaste (1400ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); Null hypothesis considered population means for the AmF toothpaste (1400ppmF) and Na MFP/NaF toothpaste (1450ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p = 0.0017, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 7.58, 95% CI 2-sided [2.88 to 12.27] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 8: Comparison: AmF Toothpaste (1400ppmF) vs NaF Toothpaste (675ppmF); Null hypothesis considered population means for AmF toothpaste (1400ppmF) and NaF toothpaste (675ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 11.97, 95% CI 2-sided [7.31 to 16.64] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 9: Comparison: AmF Toothpaste (1400ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for AmF toothpaste (1400ppmF) and placebo toothpaste (0ppmF) to be equal with respect to enamel remineralization potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 26.56, 95% CI 2-sided [21.88 to 31.24] — Statistical tests were 2-sided with a significance level of 0.05

3. Secondary Outcome: Change From Baseline in Enamel Fluoride Uptake Potential
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on the amount of fluoride (F) divided by the area of the enamel cores. The difference between treatments was calculated with respect to fluoride uptake by enamel.
Time Frame: Baseline to 14 days
Population: PP population: All randomized participants who received at least one dose of the study treatments or provided at least one significant measurement of fluoride uptake. Participants without any major protocol violations in given study treatment period were included in the PP population.
Measure: Mean (Standard Error); unit: micrograms (μg)* F/centimeters(cm)^2
Groups:
- Na MFP/NaF Toothpaste (1450ppmF): Reference toothpaste containing NaMFP/NaF (1450ppmF - 1000ppmF as NaMFP and 450ppmF as NaF)
- NaF Toothpaste (675ppmF): Toothpaste containing NaF/ silica (675ppmF)
- Placebo Toothpaste (0ppmF): Placebo: Fluoride free toothpaste
Arm/Group | NaF Toothpaste (1426ppmF) | AmF Toothpaste (1400ppmF) | Na MFP/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Number analyzed (Participants) | 56 | 57 | 58 | 59 | 59
micrograms (μg)* F/centimeters(cm)^2 | 2342.35 (123.65) | 2305.11 (123.83) | 1809.74 (121.83) | 1649.44 (121.93) | 462.95 (120.92)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426ppmF) vs AmF Toothpaste (1400ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and AmF toothpaste (1400ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p = 0.7912, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 37.24, 95% CI 2-sided [-239.62 to 314.09] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 2: Comparison: NaF Toothpaste (1426ppmF) vs Na MFP/NaF Toothpaste (1450ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and Na MFP/NaF toothpaste (1450ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p = 0.0002, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 532.61, 95% CI 2-sided [259.06 to 806.16] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 3: Comparison: NaF Toothpaste (1426ppmF) vs NaF Toothpaste (675ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and NaF toothpaste (675ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 692.91, 95% CI 2-sided [418.73 to 967.09] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 4: Comparison: NaF Toothpaste (1426ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for the NaF toothpaste (1426ppmF) and Placebo toothpaste (0ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 1879.40, 95% CI 2-sided [1605.75 to 2153.04] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 5: Comparison: AmF Toothpaste (1400ppmF) vs Na MFP/NaF Toothpaste (1450ppmF); Null hypothesis considered population means for AmF toothpaste (1400ppmF) and Na MFP/ NaF toothpaste (1450ppmF) and to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p = 0.0005, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 495.38, 95% CI 2-sided [221.09 to 769.66] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 6: Comparison: AmF Toothpaste (1400ppmF) vs NaF Toothpaste (675ppmF); Null hypothesis considered population means for AmF toothpaste (1400ppmF) and NaF toothpaste (675ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 655.67, 95% CI 2-sided [382.41 to 928.93] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 7: Comparison: AmF Toothpaste (1400ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for AmF toothpaste (1400ppmF) and placebo toothpaste (0ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 1842.16, 95% CI 2-sided [1568.73 to 2115.60] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 8: Comparison: Na MFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); Null hypothesis considered population means for the Na MFP/NaF toothpaste (1450ppmF) and NaF toothpaste (675ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p = 0.2448, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 160.30, 95% CI 2-sided [-110.58 to 431.18] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 9: Comparison: Na MFP/NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for the Na MFP/NaF toothpaste (1450ppmF) and Placebo toothpaste (0ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 1346.79, 95% CI 2-sided [1076.46 to 1617.11] — Statistical tests were 2-sided with a significance level of 0.05
Statistical Analysis 10: Comparison: NaF Toothpaste (675ppmF) vs Placebo Toothpaste (0ppmF); Null hypothesis considered population means for the NaF toothpaste (675ppmF) and Placebo toothpaste (0ppmF) to be equal with respect to enamel fluoride uptake potential; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA based on a mixed model with factors subject, treatment and period was used; Adjusted Mean Difference = 1186.49, 95% CI 2-sided [915.38 to 1457.60] — Statistical tests were 2-sided with a significance level of 0.05

ADVERSE EVENTS:
Time Frame: All AEs encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- NaMFP/ NaF Toothpaste (1450ppmF): Reference toothpaste containing NaMFP/ NaF (1450ppmF - 1000ppmF as NaMFP and 450ppmF as NaF)
Arm/Group | NaF Toothpaste (1426ppmF) | AmF Toothpaste (1400ppmF) | NaMFP/ NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF) | Overall
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57 | 0/59 | 0/59 | 0/59 | 0/65
Other Adverse Events (participants affected / at risk) | 1/57 | 5/57 | 0/59 | 3/59 | 2/59 | 10/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF Toothpaste (1426ppmF) (N=57) | AmF Toothpaste (1400ppmF) (N=57) | NaMFP/ NaF Toothpaste (1450ppmF) (N=59) | NaF Toothpaste (675ppmF) (N=59) | Placebo Toothpaste (0ppmF) (N=59) | Overall (N=65)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 2 (2) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.